CLINICAL TRIAL: NCT00235690
Title: Pharmacokinetics and Pharmacodynamics of Intravenous Colistin- Pilot Study
Brief Title: Optimizing Dosing of Colistin for Infections Resistant to All Other Antibiotics, Approved NIH Protocol Dated 12.06.07(DMID Protocol #07-0036)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 0509011; NIH
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Bacteremia; Pseudomonas Infections
MeSH Terms: conditions — Bacteremia; Pseudomonas Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- blood draws (Other): all patients enrolled will have PK blood samples obtained around a colistin dosing
  Interventions: Procedure: Blood draws; Other: Blood draw

INTERVENTIONS:
Procedure: Blood draws — PK samples obtained around a clinical dosing of colistin
Other: Blood draw — PK blood samples will be obtained around a clinical dosing of colistin

SUMMARY:
More than 80 patients at the University of Pittsburgh Medical Center have been infected with Pseudomonas aeruginosa, lacking susceptibility to all commercially available antibiotics except "colistin". This antibiotic was developed in the 1960s and preliminary pharmacokinetic studies were performed at that time. Dosing recommendations, on the basis of these pharmacokinetic studies, are listed in the drug's product information. However, there are no dosing recommendations for patients requiring renal replacement therapy (either intermittent hemodialysis or continuous venovenous hemofiltration). Furthermore, the science of antibiotic dosing ("pharmacodynamics") has changed significantly since the 1960s and it is quite possible that the dosing recommendations listed in the product information are not optimal. Furthermore, even though physicians refer to "colistin" administration, the only intravenous form of the drug is colistin methanesulfonate (CMS). CMS is converted in the body to colistin. Both CMS and colistin have different pharmacokinetic and antimicrobial activities. For this reason, we, the investigators at the University of Pittsburgh, are performing a pilot study of the pharmacokinetics of intravenous CMS/colistin in patients requiring this antibiotic for clinical purposes. Plasma concentrations will be determined around a CMS/colistin dose once the drug has reached steady state. Concentrations in pulmonary epithelial lining fluid will also be determined in patients with pneumonia. Microbiologic and clinical endpoints will be determined and will be correlated with these concentrations. The measurement of CMS and colistin levels will be determined by a laboratory in Australia which developed these assays. A submission is being made to the National Institutes of Health (NIH) for funding of a multicenter study which will address this research question with a greater sample size. The study proposed here is a pilot study in order to prove the feasibility of the research approach and to provide preliminary data for the NIH proposal.

DETAILED DESCRIPTION:
At baseline (upon signing informed consent), the following information will be collected: Demographic data - age, sex, height, weight, state of birth, underlying illnesses, underlying infection, immunosuppression, antibiotic use, laboratory results, current medication use, any other prior medical problems/history and clinical outcomes.

The research coordinator will contact the patient on days 14, 28 and 90 days after the infection to determine clinical outcome. If the patient is still an inpatient the research coordinator will visit the patient in their hospital room to evaluate the patient's health status. This visit will take about 10 minutes. If the patient has been discharged from the hospital, the patient will be contacted by telephone by the research coordinator to determine the health status, if no recent electronic medical record exists. This telephone contact will take about 10 minutes.

Blood work and microbiologic samples to be collected:

Collection of six samples of 3 mL blood on the third or fourth day of colistin therapy will occur. These samples will be collected:

* immediately pre-dose,
* at the end of the colistin infusion,
* 30 minutes after the end of the colistin infusion,
* 60 minutes after the end of the colistin infusion,
* 4 hours after the end of the colistin infusion,
* 12 hours after the end of the colistin infusion (or immediately prior to the next dose if the drug is being given every 12 hours).

Indwelling venous and arterial access lines, if already in place, will be utilized for the pharmacological study's blood draws.

Rationale: The samples will be utilized for quantification of plasma levels of colistin.

Collection of microbiologic samples within 48-96 hours of the initiation of colistin therapy. These samples are two sets of blood cultures if the patient had bacteremia, a mini-BAL for quantitative bacterial culture if the patient had pneumonia and a cerebrospinal fluid collection if the patient had Gram negative meningitis and has a cerebrospinal fluid drain in situ. Additionally, these samples will be used to determine the concentrations of colistin and CMS at the site of infection. A 3mL blood sample will be taken at the same time as these specimen collections to determine concomitant serum concentrations of colistin and CMS.

Rationale: These samples will be used to determine if there has been rapid bacteriologic clearance of infection and to determine the concentrations of drug at the site of infection.

The blood samples will be processed and stored in a -80° C freezer in a secured laboratory under the supervision of the principal investigator. These samples will then be sent to the laboratory of Drs Jian Li and Roger Nation in Melbourne, Australia, to determine the amount of colistin and CMS that reached the participant's blood following dose administration. All samples will be sent de-identified.

All samples will be analyzed to obtain the amount of colistin and CMS found in the blood. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. All samples sent outside of the UPMC facility will be de-identified. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples at UPMC will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street. All patients will be seen at the UPMC facility while they are inpatients.

Other items to be collected for study purposes:

Microbiology - the organism that caused the infection will be sub-cultured in the clinical microbiology laboratory (after the diagnosis has been obtained since the microbiology lab would otherwise destroy the culture) and provided to the investigators. All subsequent Gram negative bacterial isolates will be sub-cultured and stored for similar purposes.

An unopened vial of colistin from the same batch as used for the patient will be collected for analysis, so the actual dose of colistin can be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than 18 years of age.
* All patients will remain in the hospital for pharmacokinetic sampling.
* All subjects must be on the medication colistin as part of their standard of care.
* All individuals approached for participation shall be able to read and comprehend English.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To provide pharmacokinetic data on intravenous (IV) CMS/colistin | 5 years

SECONDARY OUTCOMES:
Determine if CMS/colistin dosing is suboptimal in ill patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Nation RL, Garonzik SM, Li J, Thamlikitkul V, Giamarellos-Bourboulis EJ, Paterson DL, Turnidge JD, Forrest A, Silveira FP. Updated US and European Dose Recommendations for Intravenous Colistin: How Do They Perform? Clin Infect Dis. 2016 Mar 1;62(5):552-558. doi: 10.1093/cid/civ964. Epub 2015 Nov 25. PMID 26607424